CLINICAL TRIAL: NCT05384964
Title: Nurses' Knowledge, Barriers and Practices in the Assessment of Delirium in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Sandra Lange, Master of Science in Nursing, MSN, Medical University of Gdansk
Other Study IDs: NKBBN/267/2022
Record Dates: First submitted 2022-05-16; First posted 2022-05-23 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Delirium; Health Knowledge, Attitudes, Practice; Critical Care Nursing
Keywords: Knowledge; Barriers; Practices; Delirium; ICU nurse; Critical care
MeSH Terms: conditions — Delirium; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire completed by ICU nurses

SUMMARY:
Delirium in intensive care patients is a complication associated with many adverse consequences. It negatively affects patient outcomes, is an independent predictor of mortality, prolongs intensive care unit (ICU) stay and causes cognitive impairment. It is estimated that delirium affects up to 80% of ICU patients. Unfortunately, delirium still remains undiagnosed in many cases. Due to the high prevalence of this complication in critically ill patients, it is important to implement an effective management protocol to prevent delirium.

Nurses' knowledge of delirium, learning about nursing practices and identifying barriers to delirium assessment, may be an important basis for early recognition and the creation of procedures for delirium prevention in the intensive care unit.

DETAILED DESCRIPTION:
The survey questionnaire is aimed at nurses working in the intensive care unit.

First, respondents are asked to answer questions on socio-demographic data. Then, two questionnaires were used to conduct the study:

1. The Nurses' Knowledge of Delirium questionnaire.

   The questionnaire consists of two parts:
   * The first part deals with questions related to the definition of delirium and the tools used to detect specific conditions.
   * In the second part, participants are asked to answer questions about delirium and its associated risk factors by ticking respectively "agree", "disagree" or "not sure" to a series of 28 statements.

   Fourteen of these statements relate to delirium, its symptoms and management, and 14 relate to risk factors for delirium.
2. Nursing Practices and Perceptions Towards Delirium in the Intensive Care Unit questionnaire.

The questionnaire consists of two parts:

* The first part consists of questions about sedation and delirium assessment.
* The second part deals with practices/opinions about delirium and its assessment, including identification of potential barriers to delirium assessment

Consents were obtained from the authors for the use of both research tools. Completion of the questionnaire is voluntary, anonymous and equivalent to giving informed consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Nurses,
* ICU staff.

Exclusion Criteria:

* Other medical staff,
* children's ICU staff,
* nurses working in other departments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will include nurses working in an adult intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Knowledge of delirium | 4 month
  Assessment of nurses' knowledge of delirium in the intensive care unit using The Nurses' Knowledge of Delirium questionnaire.
Barriers to delirium assessment | 4 month
  Identifying barriers to assessment and treatment of delirium in the intensive care unit using The Nursing Practices and Perceptions Towards Delirium in the Intensive Care Unit questionnaire.
Practices and perceptions of delirium | 4 month
  Exploring nurses' practices and perceptions of delirium in the intensive care unit using The Nursing Practices and Perceptions Towards Delirium in the Intensive Care Unit questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Wioletta Mędrzycka-Dąbrowska, Dr. Habil., Study Chair — Medical University of Gdańsk, Department of Anesthesiology Nursing & Intensive Care; Sandra Lange, MSN, Principal Investigator — Medical University of Gdańsk, Department of Internal and Pediatric Nursing
Locations (1):
- Department of Internal and Pediatric Nursing/ Department of Anesthesiology Nursing & Intensive Care, Gdansk, Gdansk/Pomorskie, Poland, Poland

REFERENCES:
- [Derived] Lange S, Medrzycka-Da Browska W, Tomaszek L, Wujtewicz M, Krupa S. Nurses' knowledge, barriers and practice in the care of patients with delirium in the intensive care unit in Poland-A cross-sectional study. Front Public Health. 2023 Mar 3;11:1119526. doi: 10.3389/fpubh.2023.1119526. eCollection 2023. PMID 36935691